CLINICAL TRIAL: NCT02267421
Title: An 8 Week Randomized Controlled Trial Assessing Home Exercise Therapy in Early Cirrhosis
Brief Title: Effects of Home Based Exercise Therapy in Early Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKPTMHLivCirHomeTraining
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home based aerobic exercise (Experimental): Home based aerobic exercise on cycle ergometer. Three times per week, 30-60 minutes per session.
  Interventions: Behavioral: Home based Aerobic exercise training
- Usual Care group (No Intervention): These patients will continue with their normal activities of daily living and will not be provided with equipment or coaching for home based exercise during the study period .

INTERVENTIONS:
Behavioral: Home based Aerobic exercise training
  Arms: Home based aerobic exercise

SUMMARY:
Individuals with Cirrhosis have been shown to have a low aerobic capacity. While supervised exercise training has been shown to be an effective intervention to remedy this, there is currently no data on home based exercise interventions in this population. This study will evaluate the effects of a home based exercise program on the aerobic capacity of enrolled early stage liver cirrhosis patients, as well as changes in quality of life, thigh muscle thickness, and thigh muscle oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

- Age >18 and less than or equal to 70 years Liver Cirrhosis Child Pugh Class A or B If required, primary or secondary Variceal prophylaxis in place

Exclusion Criteria:

- Post-liver transplantation Hepatocellular carcinoma beyond transplant criteria Active non-hepatocellular carcinoma malignancy Significant cardiac disease Hemoglobin (<80 g/L) Oxygen saturation at rest <95% Known myopathy Chronic renal failure on dialysis Physical impairment making it impossible to ride an exercise bike or treadmill Orthopedic abnormality preventing exercise training HIV infection Patient unwilling to consent to study Child Pugh class C

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in peak exercise pulmonary oxygen uptake (VO2peak). | Baseline (day 1) and Study End (8 weeks)

SECONDARY OUTCOMES:
Change in muscle mass as measured by thigh ultrasound | Baseline (day 1) and Study end (8 weeks)
Change in quality of life - Chronic Liver Disease Questionnaire | Baseline (Day 1) and Study completion (8 weeks)
Change in muscle oxygen extraction and consumption as measured by MRI | Baseline (day 1) and study completion (8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Mazankowski Heart Institute, Edmonton, Alberta, Canada

REFERENCES:
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: MedlinePlus Cirrhosis — http://www.nlm.nih.gov/medlineplus/cirrhosis.html
- See also: MedlinePlus Exercise and Physical Fitness — http://www.nlm.nih.gov/medlineplus/exerciseandphysicalfitness.html
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks